CLINICAL TRIAL: NCT03848195
Title: Hip Fracture in Individuals Under 60 Years of Age: A Prospective Multi-center Study of the Epidemiology, Treatment, Outcome and Patient Satisfaction Regarding Hip Fractures
Brief Title: Hip Fracture in Individuals Under 60 Years of Age
Acronym: HFU-60
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: University of Copenhagen (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Sebastian Strøm Rönnquist, MD, orthopaedic surgeon, PhD-student, Lund University
Other Study IDs: HFU-60
Record Dates: First submitted 2018-11-28; First posted 2019-02-20 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
Keywords: hip fractures; adult; middle-aged; DXA-scan; osteoporosis
MeSH Terms: conditions — Hip Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study prospectively analyses and describes a cohort of non-elderly hip fracture patients at four orthopaedic departments in two Scandinavian countries regarding epidemiology, treatment, Patient Reported Outcome Measures, functional outcome as well as clinical results.

DETAILED DESCRIPTION:
Hip fracture is common and well studied in the elderly population, but quite rare in the non-elderly and scarcely investigated in the literature. This prospective observational study focuses on individuals between 18 and 59 years old who have incurred a hip fracture and been treated at any of the participating orthopaedic departments in Sweden or Denmark. The study group is analysed and described at the time of the fracture and are followed during two years.

The patients' treatment follows the departments' standard rationale, there is no intervention in the study. Patients are included, after being informed and consent to participate is given, at the ward when they are admitted at the time of the fracture. The study comprises written enquiries (Patient Reported Outcome Measures, PROM) regarding hip- and global health before the fracture as well as interview and medical files and x-ray information regarding previous illness and use of medication, information about the injury, fracture type and treatment. Blood samples are used to investigate possible comorbidities and evaluate the hormonal and nutritional status and dual energy x-ray absorptiometry (DXA) is analysed with regards to reduced bone mineral density (osteopenia/-porosis). For patients with a femoral neck fracture who are treated with osteosynthesis, MRI with metal reduction is performed post-operatively and at 4 and 12 months to assess fracture healing and avascular necrosis of the femoral head.

Patients are followed up at 6 weeks by written PROM-enquiries by mail, and at 4, 12 and 24 months post-operatively with x-ray and visits in the outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Acute non-pathologic hip fracture regardless of trauma energy level or previous medical conditions.

Exclusion Criteria:

* Fracture older than four weeks.
* Not able to follow up, e.g. not living in the department area.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Among hip fracture patients treated at the participating departments, patients aged 18 to 59 years, who sustain an acute non-pathological hip fracture and are treated within four weeks, are invited to participate in the study. All patients are invited, regardless of medical, cognitive and functional pre-fracture status. The participating orthopaedic departments are part of local hospitals, treating all patients in the catchment area who seeks medical care at low (Sweden) or no cost (Denmark).
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) at the time of the fracture | Baseline
  Analysis of BMD measured by DXA-scan at the time of the fracture.
Trauma mechanism leading to the hip fracture | Baseline
  Analysis of trauma mechanism, defined as "low-energy trauma" or "not low-energy trauma", leading to the hip fracture.
Hip fracture type according to Garden classification (femoral neck fractures) and Arbeitsgemeinschaft für Osteosynthesefragen (AO)-classification (other hip fractures) | Baseline
  Analysis of the patients' hip fracture types on diagnostic radiographs.
EQ-5D | Patients are followed up during two years
  Analysis of outcome with EQ5D (PROM). A 5 dimensions, 3-levels, questionnaire regarding general health. A subscore of 1-3 for each dimension combines into a 5 digit code where lower value for each dimension indicate better outcome (total range 11111-33333).
EQ-VAS | Patients are followed up during two years
  Analysis of outcome with EQ-VAS (PROM). A visual analog scale regarding general health ranging from 0-100 where lower value indicate worse outcome.
Oxford Hip Score | Patients are followed up during two years
  Analysis of outcome with Oxford Hip Score (PROM). A 12-item, 5-levels, questionnaire on hip problems in activities of daily living. The subscores 0-4 is added to a total score for the 12 items where a higher score indicate a better outcome (total range 0-48).
VAS-pain, satisfaction, rehabilitation (VAS-psr) | Patients are followed up during two years
  Analysis of outcome with VAS-psr (PROM). Three visual analog scales (one for each dimension) regarding pain, satisfaction and rehabilitation ranging from 0-100 where lower value indicate better outcome.
New Mobility Score | Patients are followed up during two years
  Analysis of outcome with New Mobility Score (PROM). A 3-items questionnaire regarding walking ability. Each item is scored 1-3 and added into a total score where higher score indicate better outcome (total range 3-9).
Timed up and go | Patients are followed up during two years
  Analysis of outcome with timed up and go test (functional) measured in seconds. Shorter time indicates better outcome.
10 meter walking test | Patients are followed up during two years
  Analysis of outcome with 10 meter walking test (functional) measured in seconds. Shorter time indicates better outcome.
Hand grip strength | Patients are followed up during two years
  Analysis of outcome with hand grip strength (functional) measured in kg. Higher value indicates better outcome.
Complications after hip fracture surgery | Patients are followed up during two years
  Type and rate of complications after hip fracture surgery (clinical) are recorded.
Reoperations after hip fracture surgery | Patients are followed up during two years
  Type and frequency of reoperations after hip fracture surgery (clinical).
Radiological outcome after hip fracture surgery | Patients are followed up during two years
  Analysis of radiological outcome after hip fracture surgery. Radiographs are assessed according to pre-defined criteria.
Diagnosis of avascular necrosis by MRI with metal artefact reduction | Patients are followed up during two years
  Analysis of the use of MRI MARS to assess avascular necrosis of the femoral head in patients with femoral neck fracture treated with internal fixation.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Rogmark, MD, PhD, Study Director — Lund University, Skane University Hospital, Department of Orthopaedics, Sweden
Locations (4):
- Denmark (3):
  - Department of Orthopaedics, Copenhagen University Hospital Hvidovre, Hvidovre
  - Department of Orthopaedic Surgery and Traumatology, Kolding Hospital - part of Hospital Lillebaelt, Kolding
  - Department of Orthopaedic Surgery and Traumatology, Odense University Hospital, Odense
- Skane University Hospital, Department of Orthopaedics, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2018-11-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03848195/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT03848195/SAP_001.pdf